CLINICAL TRIAL: NCT04188418
Title: Efficacy and Safety of Rapid-Onset Opioids for Exertional Dyspnea in Cancer Patients
Brief Title: Fentanyl Buccal Tablet or Morphine for Exertional Dyspnea in Cancer Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-0701; NCI-2019-07529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0701 (Other: M D Anderson Cancer Center); R01CA231471 (NIH)
Record Dates: First submitted 2019-11-14; First posted 2019-12-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Fentanyl; Morphine; Exercise Test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (shuttle walk test, FBT) (Experimental): Patients complete shuttle walk test on days 1, 5, 8, 12, 15, and 19. Patients also receive FBT sublingually daily on days 6-19.
  Interventions: Drug: Fentanyl Citrate Buccal Tablet; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (shuttle walk test, morphine) (Experimental): Patients complete shuttle walk test on days 1, 5, 8, 12, 15, and 19. Patients also receive morphine PO daily on days 6-19.
  Interventions: Drug: Morphine; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (shuttle walk test, placebo) (Active Comparator): Patients complete shuttle walk test on days 1, 5, 8, 12, 15, and 19. Patients also receive placebo (sublingually or PO) daily on days 6-19.
  Interventions: Other: Physical Performance Testing; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Fentanyl Citrate Buccal Tablet — Given transmucosally
  Other Names: Fentora
  Arms: Group I (shuttle walk test, FBT)
Drug: Morphine — Given PO
  Arms: Group II (shuttle walk test, morphine)
Other: Physical Performance Testing — Complete shuttle walk test
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Placebo Administration — Given PO
  Arms: Group III (shuttle walk test, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies fentanyl buccal tablet or morphine to see how well it works compared to a placebo in controlling shortness of breath during or after physical activity in cancer patients. Fentanyl sublingual tablet and morphine are opioids normally used to control pain that may also help to prevent or control shortness of breath during or after physical activity in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the effect of prophylactic fentanyl buccal tablet (FBT), morphine sulfate, and placebo on the increase in the intensity of exertional dyspnea (0-10 point modified Borg scale) measured before versus at the end of a shuttle walk test (SWT).

SECONDARY OBJECTIVES:

I. To compare the effects of prophylactic FBT, morphine sulfate, and placebo on SWT distance and dyspnea unpleasantness, average daily dyspnea (intensity and unpleasantness, oxygen cost diagram), personalized daily activity (ability to complete activity), personalized dyspnea response, symptom burden (Edmonton Symptom Assessment System [ESAS]), quality of life (EuroQol-5 Dimension-5 Level [EQ-5D-5L]), and dyspnea severity and functional impairment based on the Patient Reported Outcomes Measurement Information System (PROMIS) dyspnea instruments.

II. To explore the effects of prophylactic FBT, morphine sulfate, and placebo on neurocognitive function, addictive potential (Drug Effects Questionnaire), adverse effects (Common Terminology Criteria for Adverse Events [CTCAE], Patient-Reported Outcomes version of CTCAE [PRO-CTCAE]), and pattern of opioid use.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients complete shuttle walk test on days 1, 5, 8, 12, 15, and 19. Patients also receive FBT sublingually daily on days 6-19.

GROUP II: Patients complete shuttle walk test on days 1, 5, 8, 12, 15, and 19. Patients also receive morphine orally (PO) daily on days 6-19.

GROUP III: Patients complete shuttle walk test on days 1, 5, 8, 12, 15, and 19. Patients also receive placebo (sublingually or PO) daily on days 6-19.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer with evidence of active disease
2. Dyspnea on exertion with an average intensity level ≥4/10 on a modified Borg scale
3. Outpatient at participating centers
4. Ambulatory and able to walk, with or without walking aid
5. On strong opioids with morphine equivalent daily dose (MEDD) of 60-400 mg for ≥1 wk (i.e. at least 4 out of 7 days), with stable (i.e. ±30%) regular dose over the last 3 d
6. Karnofsky performance status ≥40%
7. Age ≥18 yrs
8. Able to complete study assessments
9. Able to speak English or Spanish
10. Reside within 65 miles of participating centers or expected to visit MD Anderson in person at least once a month

Exclusion Criteria:

1. Dyspnea at rest ≥7/10 on modified Borg scale at enrollment
2. Supplemental oxygen requirement >6 L/min
3. Delirium (i.e. Memorial Delirium Assessment Scale ≥13)
4. History of unstable angina or myocardial infarction 1 mo prior to enrollment
5. Hemodynamic instability requiring hospitalization
6. History of substance use disorder or abnormal urinary drug screen within the past year, or at risk of opioid abuse as determined by Screener and Opioid Assessment for Patients with Pain (SOAPP14) ≥7
7. History of or known allergy to fentanyl or morphine sulfate
8. Using scheduled benzodiazepines at the time of enrollment and cannot stop during the study
9. Severe anemia (Hb <7 g/L) if documented in the last month and not corrected prior to study enrollment*
10. Bilirubin ≥5x upper limit of normal if documented in the last month and not lowered to <5x normal prior to enrollment*
11. Diagnosis of acute pulmonary embolism within past 2 wks
12. Diagnosis of pulmonary hypertension
13. Diagnosis of malignant pleural effusion with therapeutic thoracentesis expected in the next 2 wks
14. Currently pregnant or breastfeeding
15. Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in modified Borg scale dyspnea intensity before and after the Shuttle Walk Test (SWT) | Days 5, 8, 12, 15, and 19
  Will first determine whether the three treatment groups are different; if so, will test the three pairwise comparisons with intention-to-treat analyses. Repeated-measures analysis of variance (ANOVA) will be implemented using linear mixed effects models with the difference in intervention period SWT modified Borg scale dyspnea intensity before and after SWT as the response variable and the treatment group and observation period SWT measures as predictor variables.

SECONDARY OUTCOMES:
SWT distance | Days 5, 8, 12, 15, and 19
  Will be analyzed using linear mixed effects models similar to the primary analysis.
Dyspnea unpleasantness | Days 5, 8, 12, 15, and 19
  Will be analyzed using linear mixed effects models similar to the primary analysis.
Daily dyspnea intensity and unpleasantness | Days 1-19
  Will be analyzed using linear mixed effects models similar to the primary analysis.
Personalized daily activity | Days 1-4, 6-7, 9-11, 13-14, and 16-18
  Will be analyzed using linear mixed effects models similar to the primary analysis.
Oxygen cost diagram | Days 1-19
  Will be analyzed using linear mixed effects models similar to the primary analysis.
Symptom burden Questionnaires | Days 1-19
  Will be measured by the Edmonton Symptom Assessment System and analyzed using linear mixed effects models similar to the primary analysis.
Quality of life Questionnaires | Days 1-19
  Will be measured by the EuroQol-5 Dimension-5 Level Questionnaire and analyzed using linear mixed effects models similar to the primary analysis.
Neurocognitive function | Up to day 19
  Will perform paired t-test or ANOVA if the data are normally distributed and the Wilcoxon rank-sum test or Kruskal-Wallis if the data are non-normal.
Addictive potential | Up to day 19
  Will be measured by the Drug Effects Questionnaire. Will perform paired t-test or ANOVA if the data are normally distributed and the Wilcoxon rank-sum test or Kruskal-Wallis if the data are non-normal.
Frequency, severity, and interference of adverse effects | Up to day 19
  Will be measured by the Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE). Will perform paired t-test or ANOVA if the data are normally distributed and the Wilcoxon rank-sum test or Kruskal-Wallis if the data are non-normal.
Total opioid dose | Up to day 19
  Will perform paired t-test or ANOVA if the data are normally distributed and the Wilcoxon rank-sum test or Kruskal-Wallis if the data are non-normal.
Number of rescue doses per day | Up to day 19
  Will perform paired t-test or ANOVA if the data are normally distributed and the Wilcoxon rank-sum test or Kruskal-Wallis if the data are non-normal.
Dyspnea severity and functional impairment | Day 1, 5, 12, 19
  Will be measured using the Patient Reported Outcomes Measurement Information System (PROMIS) dyspnea instruments.

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Pacheco S, Nguyen L, Jennings K, de la Cruz V, Stanton P, Laureano R, Ontai A, Mahler D, Bruera E. Efficacy of fentanyl buccal tablet and morphine for exertional dyspnoea in patients with cancer: a double-blind, placebo-controlled, randomised clinical trial. Thorax. 2025 Oct 20:thorax-2025-222970. doi: 10.1136/thorax-2025-222970. Online ahead of print. PMID 41115797
- See also: M D Anderson Cancer Center — http://www.mdanderson.org